CLINICAL TRIAL: NCT00235807
Title: Multi-Site Randomized Clinical Study of Tinnitus Treatment Methods
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Henry, James - Principal Investigator, Department of Veterans Affairs
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C3214R
Record Dates: First submitted 2005-10-06; First posted 2005-10-10 (Estimated); Last update posted 2011-03-24 (Estimated); Status verified 2011-03

CONDITIONS: Tinnitus
Keywords: Audiology; Rehabilitation; Tinnitus
MeSH Terms: conditions — Tinnitus

ARMS (3):
- 1 (Other): should contain an explanation of the nature of the study group (e.g., those with a condition and those without a condition; those with an exposure and those without an exposure).
  Interventions: Procedure: Tinnitus Masking
- 2 (Other): should contain an explanation of the nature of the study group (e.g., those with a condition and those without a condition; those with an exposure and those without an exposure).
  Interventions: Procedure: Tinnitus Retraining Therapy (TRT)
- 3 (Other): should contain an explanation of the nature of the study group (e.g., those with a condition and those without a condition; those with an exposure and those without an exposure).
  Interventions: Procedure: Tinnitus Education (TED)

INTERVENTIONS:
Procedure: Tinnitus Masking — Sound therapy with Tinnitus Masking is intended to produce immediate relief from the discomfort caused by tinnitus (Vernon, 1977; 1987; Vernon, 1988). If maskers or combination units are used, the masking sound can be set at any level the patient chooses to attain maximum relief. Relief using masking noise can be accomplished using the external sound of the masker, which is generally a more acceptable sound than the tinnitus.
  Arms: 1
Procedure: Tinnitus Retraining Therapy (TRT) — The TRT procedure adheres as closely as possible to the methodology described by Dr. Pawel Jastreboff. For TRT, sound therapy is used to facilitate long-term habituation to tinnitus (Jastreboff, 1999b).
  Arms: 2
Procedure: Tinnitus Education (TED) — TED represents tinnitus treatment that would typically be provided by audiologists using hearing aids and counseling (although for this study the counseling has been structured and expanded to be equivalent in length to the other two groups).
  Arms: 3

SUMMARY:
The purpose of this multi-site randomized clinical study was to assess treatment outcomes for three forms of tinnitus treatment: Tinnitus Retraining Therapy (TRT), Tinnitus Masking, and Tinnitus Education (TED). There were four study sites: VAMC Audiology Clinics at Bay Pines, FL; Portland, OR; Seattle, WA; and San Diego, CA. Thirty-six subjects (Veterans) were enrolled into treatment at each site - 12 into each treatment group. Each subject received 18 months of treatment. Treatment appointments and outcome questionnaires occurred at 0, 3, 6, 12, and 18 months. Qualified subjects were initially randomized to one of the treatment groups or to a 6-month Waiting List group. Those in the Waiting List group completed outcome questionnaires at 3 and 6 months, and were randomized into one of the three treatment groups. They then received 18 months of treatment as above.

DETAILED DESCRIPTION:
Although tinnitus is especially problematic for Veterans, the DVA has no established protocol for tinnitus rehabilitation. We recently completed a randomized clinical trial to evaluate the efficacy of tinnitus treatment for veterans. Tinnitus Masking and Tinnitus Retraining Therapy (TRT) were both shown to be effective for the majority of Veterans treated with these methods by expert tinnitus clinicians. The objective of the present study was to determine if the same level of treatment efficacy observed in the previous study could be obtained by typical VA audiologists in their clinical environment. In addition, a third group was added, called Tinnitus Education (TED), which served as a control group for nonspecific effects of treatment using a standardized protocol of hearing aids and education.

Veterans with clinically significant tinnitus were recruited to receive treatment with Masking, TRT, or TED in Audiology Clinics at the Bay Pines, Portland, San Diego, and Seattle VAMCs. There were three Treatment Audiologists at each of the sites, one for each of the three treatment methods. Each method uses a variation of sound therapy and of educational counseling. Sound therapy involves the use of wearable ear-level devices, including sound generators (maskers), hearing aids, or combination devices (hearing aid and masker combined). Only the TED group was restricted to the use of hearing aids only (note: TED subjects who did not require hearing aids were the only subjects in this study who did not receive ear-level devices). TRT uses a structured counseling protocol that teaches concepts that are unique to TRT. The Masking protocol has been created to match the TRT counseling with respect to comparable formatting and length of counseling sessions, but containing information specific to the concepts of Masking. The TED counseling protocol is similarly matched in format and length, but the information conveyed is of a more generic nature (general audiologic counseling information). Assessment of outcomes utilized questionnaires that were administered at intervals before, during, and after the 18 months of treatment.

Potential participants at all sites were telephone-screened by the Project Audiologist in Portland to determine if the tinnitus is a clinically significant problem warranting 18 months of treatment. Veterans who passed the screening were scheduled to meet with the Research Coordinator (RC) at the respective study site. At this first visit, Veterans were consented, completed questionnaires, and were then informed as to their group placement. Per a randomization schedule, they were placed into one of the three treatment groups, or into the 6-month waiting list group (with treatment starting 6 months later). At the initial evaluation with the respective Treatment Audiologist, a tinnitus verbal interview was administered, hearing and tinnitus testing were performed, and ear mold impressions were taken to order the custom ear-level devices. The Veteran returned approximately 3-4 weeks later to be fitted with the devices and to receive the counseling/education that initiates treatment. Subjects returned for follow-up treatment at 3, 6, 12 and 18 months. At the follow-up appointments, the RC collected and checked the questionnaires, and the Treatment Audiologist administered the follow-up verbal interview and repeated the counseling protocol.

ELIGIBILITY:
Inclusion Criteria:

* Veterans with a) clinically significant tinnitus, and b) no significant language barrier.

Exclusion Criteria:

* Any medical conditions that would interfere with study participation (e.g., medically or surgically treatable otologic disease; end-stage renal, pulmonary, or cardiovascular disease; patients undergoing chemotherapy or radiation treatment; and patients with severe psychiatric disorders). Subjects must be free from such conditions and will be required to: (1) be between the ages of 2180; and (2) have a weighted error score of 10 or less on the Blessed Orientation-Memory Concentration Test.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2004-06; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Tinnitus Handicap Inventory (THI) | Baseline, 3 months, 6 months, 12 months, 18 months

SECONDARY OUTCOMES:
Tinnitus Severity Index (TSI) | Baseline, 3 months, 6 months, 12 months, 18 months

CONTACTS AND LOCATIONS:
Overall Officials: James Henry, PhD, Principal Investigator — VA Medical Center, Portland
Locations (1):
- VA Medical Center, Portland, Portland, Oregon, United States

REFERENCES:
- See also: Click here for more information about this study: Multi-Site Randomized Clinical Study of Tinnitus Treatment Methods — http://www.ncrar.research.va.gov/